CLINICAL TRIAL: NCT03581643
Title: Validation of the Montreal Cognitive Assessment in Patients With Mild and Major Neurocognitive Disorder
Acronym: MoCA-Valid
Status: Completed | Type: Observational
Sponsor: Andreas Monsch (Other)
Responsible Party: Sponsor-Investigator, Andreas Monsch, Professor of Psychology, Head Memory Clinic, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: MoCA-Valid
Record Dates: First submitted 2018-05-30; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Montreal Cognitive Assessment; Sensitivity; Specificity; Validation Study
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of our study is to investigate the specificity, the sensitivity, and the overall diagnostic accuracy of the MoCA for mild and major NCD in a German-speaking population.

Secondary aims are: (1) to study the MoCA performance in different patient groups and (2) to compare the diagnostic properties of the MoCA with the ones of the MMSE (i.e., the current reference standard for screening of MCI).

DETAILED DESCRIPTION:
Due to the demographical development, age-related diseases will drastically increase over the next decades. To face this healthcare challenge, early and accurate identification of cognitive impairment is crucial. The early detection of cognitive decline requires a tool that is short, easy to administer and interpret, and has high diagnostic accuracy. Currently, a widely used instrument is the Mini-Mental State Examination (MMSE). However, the MMSE sensitivity is poor when identifying individuals with MCI, and it lacks meaningful assessment of executive functions. The Montreal Cognitive Assessment (MoCA) has been developed to address these weaknesses. It has demonstrated better diagnostic accuracy in patients with MCI, has less ceiling effect, and a higher test-retest-reliability. In addition, the MoCA better captures the cognitive domains proposed in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

In 2018, the investigators generated demographically adjusted normative values for the German version of the MoCA in cognitively healthy individuals. However, these normative data alone are not suitable to determine the exact diagnostic accuracy. Therefore, the investigators aim to analyze data from patients with cognitive disorders to validate the German version of the MoCA.

Validation studies for the MoCA have been performed in various languages and different etiologies, mainly in patients with MCI and AD. However, when applying the MoCA in a clinical routine setting, the patient population is more heterogeneous and different etiologies may lead to deficits in characteristic cognitive domains. Therefore, patients with diseases other than AD may perform differently on items of the MoCA. This might translate into differences regarding the optimal cut-off score to detect possible cognitive impairment. Thus, when solely relying on a cut-off score that has been validated in a population of AD patients, patients with other diseases leading to cognitive impairment may be missed.

The investigators therefore aim to establish the diagnostic accuracy of the MoCA when applied in a clinically diverse patient sample, namely, a sample that is seen in a typical Memory Clinic. In a first step, the diagnostic properties of the MoCA will be investigated by differentiating between healthy controls and all patients with mild and major neurocognitive disorders (NCD). In a second step, healthy controls will be compared separately to patients with mild NCD and to patients with major NCD. The investigators further aim to investigate the aptness of the MoCA for differential diagnostic. The MoCA performance of different diagnostic patient groups will be compared. Investigating the presence or absence of deficits per subitem in each patient group may reveal if different etiologies lead to characteristic MoCA profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Education ≥ 7 years.
* Fluency in the German language.
* Completed neuropsychological assessment.

Exclusion Criteria:

* Severe sensory or motor impairment interfering with cognitive testing.
* Documented refusal of the use of health-related personal data.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing the routinely held neuropsychological assessments in the Memory Clinic, University Center for Medicine of Aging, Felix Platter Hospital in Basel, Switzerland.
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) total score | Administered once at baseline
  Performance on the MoCA (0-30; higher score indicates better performance)

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) total score | Administered once at baseline
  Performance on the MMSE (0-30; higher score indicates better performance)
Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB) | Administered once at baseline
  CERAD-NAB total score (0-120; higher score indicates better performance)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Monsch, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Memory Clinic, University Center for Medicine of Aging, Felix Platter Hospital Basel, Basel, Canton of Basel-City, Switzerland